CLINICAL TRIAL: NCT00829933
Title: A Randomized Dose-ranging Controlled Trial of DU-176b Versus Warfarin Potassium in Patients With Non-valvular Atrial Fibrillation
Brief Title: Late Phase 2 Study of DU-176b in Patients With Non-Valvular Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DU176b-C-J225
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2015-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Factor Xa inhibition
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban; Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): DU-176b low dose
  Interventions: Drug: DU-176b tablets
- 2 (Experimental): DU-176b intermediate dose
  Interventions: Drug: DU-176b tablets
- 3 (Experimental): DU-176b high dose
  Interventions: Drug: DU-176b tablets
- 4 (Active Comparator): Warfarin
  Interventions: Drug: Warfarin potassium tablets

INTERVENTIONS:
Drug: DU-176b tablets — DU-176b tablets taken once daily for up to 12 weeks
  Arms: 1; 2; 3
Drug: Warfarin potassium tablets — Warfarin potassium tablets taken once daily for up to 12 weeks
  Arms: 4

SUMMARY:
The primary objective of this study is to compare the incidence of hemorrhagic events in patients treated for non-valvular atrial fibrillation with DU-176b at each dose level versus warfarin potassium (warfarin). The secondary objective includes between-group comparisons with regard to incidence of thromboembolic events, pharmacodynamic parameters, and biomarkers for the efficacy evaluation, as well as incidence of adverse events and adverse reaction for the safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-valvular atrial fibrillation who meet all of the following requirements will be considered for admission to the study:

  * Age≧20years
  * Atrial fibrillation confirmed by at least 2 electrocardiographic(ECG) tracings taken at an interval of ≧1week during the year before enrollment
* Presence of any (at least )one of the following risk factors for embolism:

  * Hypertension
  * Diabetes mellitus
  * Congestive heart failure
  * Previous transient ischemic attack (TIA) or cerebral infarction (more than 30 days before giving informed consent )
  * Age≧75 years
  * At time of giving informed consent.
  * To be confirmed on ECG charts, etc.

Exclusion Criteria:

* Presence of any of the following conditions with increased risk of hemorrhage:

  * History of intracranial, intraocular (excluding bleeding beneath the bulbar conjunctiva ), intrathecal, retroperitoneal, or non-traumatic intraarticular hemorrhage
  * History of gastrointestinal hemorrhage during the year before giving informed consent
  * History of peptic ulcers during the 90 days before giving informed consent
  * Surgical treatment or trauma requiring hospitalization during the 30 days before giving informed consent
  * Hemoglobin level <10 g/dL platelet count <10 ×10000 /μL at screening examinations
  * Active hemorrhage* present at giving informed consent or at enrollment
  * Any invasive therapeutic or diagnostic procedure (e.g., surgery, tissue, biopsy, and tooth extraction) scheduled during the period from the time of informed consent until completion of the trial treatment.
  * Any congenital hemorrhagic disease
* History of cerebral infarction or TIA within 30 days before giving informed consent
* Current treatment with any anticoagulant(other than warfarin)
* Concurrent rheumatic valvular disease
* History of valvular surgery
* Concurrent infectious endocarditis
* Concurrent cardiac myxoma
* Confirmed left ventricular or left atrial thrombosis
* Any congenital condition with a tendency toward thrombosis
* Electrical or pharmacological defibrillation scheduled during the trial treatment
* Uncontrolled hypertension (persistently high systolic ［>160mmHg］or diastolic [>100mmHg] pressure)
* Uncontrolled diabetes mellitus
* Renal or hepatic dysfunction (as defined below ), confirmed at screening examinations

  * Serum creatinine>1.5mg/dL
  * AST(GOT)or ALT(GPT)≧twice the upper limit of the reference range
  * Total bilirubin ≧twice the upper limit of the reference range
* Current antiplatelet therapy for any concomitant illness that may be aggravated after discontinuation of the therapy.
* Any concurrent severe cardiac disease
* Known allergy to warfarin or any condition contraindicating its use
* Inability to discontinue current treatment with vitamin K
* Confirmed or potential pregnancy, wish to become pregnant during the study period, or current breast feeding
* Previous treatment with DU-176b
* Participation in a trial of any other drug during the 6 month before giving informed consent
* Any other condition that disqualifies the patient for the study in the opinion of the investigator/subinvestigator *This includes ecchymosis identified as at least one hematoma sized ≧5 cm in longer diameter, macroscopic hematuria, and microscopic hematuria defined as a ≧2+test or a 1+ test for occult blood with a urine sediment containing ≧10 red cells per high-power field (except for a 2+ occult blood test persisting for 1 year before giving informed consent).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Groups:
- DU-176b Low Dose 30mg; DU-176b Intermediate Dose 45mg; DU-176b High Dose 60mg: DU-176b tablets:
  DU-176b tablets taken once daily for 12 weeks
- Warfarin: Warfarin potassium tablets:
  Warfarin potassium tablets taken once daily for 12 weeks while adjusting dose
Period: Overall Study
Arm/Group | DU-176b Low Dose 30mg | DU-176b Intermediate Dose 45mg | DU-176b High Dose 60mg | Warfarin
Started | 135 | 135 | 132 | 134
Baseline Analysis Population | 131 | 134 | 131 | 129
Completed | 121 | 122 | 119 | 120
Not Completed | 14 | 13 | 13 | 14
Not completed — Adverse Event | 2 | 3 | 2 | 1
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Physician Decision | 5 | 7 | 8 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 2 | 1 | 0 | 0
Not completed — withdrew before treatment started | 5 | 1 | 2 | 9

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population is based on Full Analysis Set. FAS defined as all subjects enrolled in study, but excluded those who had GCP violations, who did not receive any dose of study drug, or who did not have atrial fibrillation confirmed by ECG performed at least twice within a 1-week or longer interval within 1 year before registration
Groups:
- DU-176b Low Dose 30mg; DU-176b Intermediate Dose 45mg; DU-176b High Dose 60mg: DU-176b tablets taken once daily for 12 weeks
- Warfarin: Warfarin potassium tablets taken once daily for 12 weeks while adjusting dose
- Total: Total of all reporting groups
Arm/Group | DU-176b Low Dose 30mg | DU-176b Intermediate Dose 45mg | DU-176b High Dose 60mg | Warfarin | Total
Number analyzed (Participants) | 131 | 134 | 131 | 129 | 525
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (7.5) | 69.5 (8.8) | 68.4 (8.2) | 68.8 (8.2) | 69.0 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 24 | 22 | 92
  Male | 110 | 109 | 107 | 107 | 433
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 131 | 134 | 131 | 129 | 525
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 131 | 134 | 131 | 129 | 525

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Bleeding Events (Major Bleeding, Clinically Relevant Non-major Bleeding and Minor Bleeding ) Identified During the Period From the Entry Into the Treatment Period Until Completion or Termination of the Treatment.
Description: The primary endpoint was the incidence of bleeding events (major bleeding, clinically relevant non-major bleeding, or minor bleeding) that occurred during the treatment period.
Time Frame: 12 weeks
Population: Primary endpoint analyzed for subjects who proceeded to treatment period in FAS.
Measure: Number (95% Confidence Interval); unit: percent of subjects with bleeding event
Arm/Group | DU-176b Low Dose 30mg | DU-176b Intermediate Dose 45mg | DU-176b High Dose 60mg | Warfarin
Number analyzed (Participants) | 130 | 134 | 130 | 125
percent of subjects with bleeding event | 18.5 [12.7 to 26.0] | 22.4 [16.2 to 30.2] | 27.7 [20.7 to 35.9] | 20.0 [13.9 to 27.9]
Statistical Analysis 1: Comparison: DU-176b Low Dose 30mg vs DU-176b Intermediate Dose 45mg; For the incidence of bleeding events, paired comparison between the DU-176b groups was performed using the χ2 test; Test type: Superiority or Other; p = 0.429, Chi-squared
Statistical Analysis 2: Comparison: DU-176b Low Dose 30mg vs DU-176b High Dose 60mg; Test type: Superiority or Other; p = 0.077, Chi-squared
Statistical Analysis 3: Comparison: DU-176b Low Dose 30mg vs Warfarin; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); Cox Proportional Hazard = -1.5, 95% CI 2-sided [-11.2 to 8.1]
Statistical Analysis 4: Comparison: DU-176b Intermediate Dose 45mg vs DU-176b High Dose 60mg; Test type: Superiority or Other; p = 0.320, Chi-squared
Statistical Analysis 5: Comparison: DU-176b Intermediate Dose 45mg vs Warfarin; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); Cox Proportional Hazard = 2.4, 95% CI 2-sided [-7.6 to 12.3]
Statistical Analysis 6: Comparison: DU-176b High Dose 60mg vs Warfarin; Test type: Superiority or Other; Wilcoxon (Mann-Whitney); Cox Proportional Hazard = 7.7, 95% CI 2-sided [-2.7 to 18.1]

2. Secondary Outcome: Incidence of Thromboembolic Events (Cerebral Infarction and Systemic Embolism) Identified During the Period From the Entry to the Treatment Period Until Completion or Termination of the Treatment.
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Incidence of Adverse Events and Adverse Reactions Identified During the Period From the Entry to the Treatment Period Until Completion or Termination of the Treatment
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Pharmacodynamic Parameters (PT, PT-INR, and APTT)
Description: PT - prothrombin time INR - International Normalized Ratio APTT - Activated Partial Thromboplastin time
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Plasma DU-176 Concentration
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Pharmacodynamic Biomarkers (F1+2, TAT, and D-dimer )
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | DU-176b Low Dose 30mg | DU-176b Intermediate Dose 45mg | DU-176b High Dose 60mg | Warfarin
Serious Adverse Events (participants affected / at risk) | 4/130 | 2/134 | 2/130 | 7/125
Other Adverse Events (participants affected / at risk) | 85/130 | 103/134 | 103/130 | 88/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b Low Dose 30mg (N=130) | DU-176b Intermediate Dose 45mg (N=134) | DU-176b High Dose 60mg (N=130) | Warfarin (N=125)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DU-176b Low Dose 30mg (N=130) | DU-176b Intermediate Dose 45mg (N=134) | DU-176b High Dose 60mg (N=130) | Warfarin (N=125)
nasopharyngitis (Infections and infestations) | 19 (19) | 25 (27) | 14 (15) | 18 (19)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (14) | 16 (17) | 6 (7)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 7 (8) | 6 (7) | 8 (12) | 6 (16)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 8 (8) | 4 (4) | 2 (2)
Blood triglycerides increased (Investigations) | 1 (1) | 5 (5) | 5 (5) | 9 (10)
Gamma-glutamyltransferase increased (Investigations) | 7 (7) | 8 (8) | 7 (7) | 4 (4)
glucose urine present (Investigations) | 5 (6) | 9 (10) | 6 (6) | 7 (8)
glood urine present (Investigations) | 17 (19) | 24 (26) | 30 (33) | 18 (20)
protein urine present (Investigations) | 3 (3) | 6 (6) | 3 (3) | 8 (8)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 4 (6) | 3 (3) | 5 (5) | 5 (5)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 4 (6) | 3 (3) | 5 (5) | 5 (5)
Alanine aminotransferase increased (Investigations) | 5 (5) | 5 (5) | 4 (4) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2) | 4 (4) | 2 (2)
Eosinophil count increased (Investigations) | 1 (1) | 3 (3) | 4 (4) | 3 (3)
Platelet count decreased (Investigations) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish the results of the Study at any time without the prior written approval of Sponsor.